CLINICAL TRIAL: NCT03428529
Title: Estudo Randomizado de Fase II Com Capecitabina Versus 5-Fluorouracil/Leucovorin em Bolus Associados à Radioterapia no Tratamento Neoadjuvante de câncer de Reto Localmente avançado: INCAGI004.
Brief Title: Capecitabine Versus Bolus 5-Fu Associated to Radiotherapy as Neoadjuvant Treatment for Rectal Cancer.
Acronym: INCAGI004
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Principal Investigator, Rodrigo Otavio de Castro Araujo, Dr. Rodrigo Otavio de Castro Araujo, Instituto Nacional de Cancer, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP INCA 83/10
Record Dates: First submitted 2018-02-05; First posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Rectal Neoplasm Malignant
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Fluorouracil

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capecitabine (Experimental): Neoadjuvant capecitabine plus RT
  Interventions: Drug: Capecitabine Oral Product
- 5-Flourouracil (Active Comparator): Neoadjuvant 5-Fluorouracil plus RT
  Interventions: Drug: 5Fluorouracil

INTERVENTIONS:
Drug: Capecitabine Oral Product — Neoadjuvant Capecitabine concomitant to external beam radiotherapy
  Other Names: Xeloda
  Arms: Capecitabine
Drug: 5Fluorouracil — Neoadjuvant bolus 5-Fluorouracil concomitante to external beam radiotherapy
  Other Names: 5-Fu
  Arms: 5-Flourouracil

SUMMARY:
A randomized two-arm study comparing preoperative CRT using oral capecitabine versus bolus 5-FU/LV concomitant to external beam radiation (50.5 Gy/28 fractions) for locally advanced rectal cancer. Main outcome was clinical response assessed using MRI and endorectal US 6-8 weeks after CRT. Secondary endpoints were pathological response, adverse effects, sphyncter preservation, quality of life, OS and DFS.

DETAILED DESCRIPTION:
Patients harbouring rectal adenocarcinoma T3-4 or N>0 M0 within 10 cm to anal verge were randomized in two treatment arms: (1) capecitabina orally 825mg/m2 bid. 5 days a week for 5 weeks and (2) bolus intravenous 5-FU/LV 350mg/m2/20 mg/m2 D1-D5 on the first and fifth weeks, both combined to pelvic radiotherapy, total dose 50.4 Gy in 28 fractions. Clinical stage before and after CRT was determined using pelvic Magnetic Resonance Imaging (MRI), endorectal ultrasonography (ERUS) and chest, abdominal and pelvic Computer Tomography. Surgery was planned 6 to 8 weeks after CRT. Sphincter preservation was always considered when negative margins were possible. Pathological assessment included stage (TNM 7th Ed.) and Mandard's Tumor Regression Grade (TRG). QOL questionnaires QLQ-C30 and CR38 were completed by patients before and after CRT, after surgery and during follow-up.

ELIGIBILITY:
Inclusion Criteria:

Patients with histologically proven locally advanced rectal cancer (cT3-4 or positive regional lymph node) on endorectal ultrasonography (EUS) or pelvic Magnetic Resonance Imaging (MRI) were qualified for this study. Distance from anal verge (AV) should not exceed 10 cm measured with rigid proctoscopy. Thorax and abdominal computer tomography (CT) exams were taken to rule out distant metastasis. Performance Status ECOG 0-1.

Exclusion Criteria:

Previous treatment for rectal cancer (RT, chemotherapy or surgical resection). Previous diagnosis of other cancers except nonmelanoma skin cancer. Uncontrolled comorbities including heart failure and miocardial infarction in the previous 6 months. Hepatic insufficiency and renal failure. Pregnancy. Serious neurologic or psyquiatric disturbances that could affect comprehension of informed consent.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2011-01-12 (Actual); Primary Completion 2016-10-13 (Actual); Study Completion 2016-12-13 (Actual)

PRIMARY OUTCOMES:
Clinical downstaging | 6-8 weeks after CRT
  Clinical downstaging after neoadjuvant treatment

SECONDARY OUTCOMES:
Pathological downstaging | 8 weeks after CRT
  Patholgical downstaging after neoadjuvant treatment

IPD SHARING:
Plan to Share IPD: No
IPD could be shared if requested after IRB approval.

REFERENCES:
- [Background] Saif MW, Hashmi S, Zelterman D, Almhanna K, Kim R. Capecitabine vs continuous infusion 5-FU in neoadjuvant treatment of rectal cancer. A retrospective review. Int J Colorectal Dis. 2008 Feb;23(2):139-45. doi: 10.1007/s00384-007-0382-z. Epub 2007 Oct 2. PMID 17909820
- [Background] Wolff HA, Conradi LC, Beissbarth T, Leha A, Hohenberger W, Merkel S, Fietkau R, Raab HR, Tschmelitsch J, Hess CF, Becker H, Wittekind C, Sauer R, Rodel C, Liersch T; German Rectal Cancer Study Group. Gender affects acute organ toxicity during radiochemotherapy for rectal cancer: long-term results of the German CAO/ARO/AIO-94 phase III trial. Radiother Oncol. 2013 Jul;108(1):48-54. doi: 10.1016/j.radonc.2013.05.009. Epub 2013 Jun 11. PMID 23768685
- [Background] Sawada N, Ishikawa T, Sekiguchi F, Tanaka Y, Ishitsuka H. X-ray irradiation induces thymidine phosphorylase and enhances the efficacy of capecitabine (Xeloda) in human cancer xenografts. Clin Cancer Res. 1999 Oct;5(10):2948-53. PMID 10537364
- [Background] Schuller J, Cassidy J, Dumont E, Roos B, Durston S, Banken L, Utoh M, Mori K, Weidekamm E, Reigner B. Preferential activation of capecitabine in tumor following oral administration to colorectal cancer patients. Cancer Chemother Pharmacol. 2000;45(4):291-7. doi: 10.1007/s002800050043. PMID 10755317
- [Background] Suarez J, Vera R, Balen E, Gomez M, Arias F, Lera JM, Herrera J, Zazpe C. Pathologic response assessed by Mandard grade is a better prognostic factor than down staging for disease-free survival after preoperative radiochemotherapy for advanced rectal cancer. Colorectal Dis. 2008 Jul;10(6):563-8. doi: 10.1111/j.1463-1318.2007.01424.x. Epub 2007 Dec 7. PMID 18070184
- [Background] Tulchinsky H, Shmueli E, Figer A, Klausner JM, Rabau M. An interval >7 weeks between neoadjuvant therapy and surgery improves pathologic complete response and disease-free survival in patients with locally advanced rectal cancer. Ann Surg Oncol. 2008 Oct;15(10):2661-7. doi: 10.1245/s10434-008-9892-3. Epub 2008 Apr 4. PMID 18389322
- [Background] Bosset JF, Collette L, Calais G, Mineur L, Maingon P, Radosevic-Jelic L, Daban A, Bardet E, Beny A, Ollier JC; EORTC Radiotherapy Group Trial 22921. Chemotherapy with preoperative radiotherapy in rectal cancer. N Engl J Med. 2006 Sep 14;355(11):1114-23. doi: 10.1056/NEJMoa060829. PMID 16971718
- [Result] Kim JS, Kim JS, Cho MJ, Yoon WH, Song KS. Comparison of the efficacy of oral capecitabine versus bolus 5-FU in preoperative radiotherapy of locally advanced rectal cancer. J Korean Med Sci. 2006 Feb;21(1):52-7. doi: 10.3346/jkms.2006.21.1.52. PMID 16479065
- [Result] Saif MW. Capecitabine versus continuous-infusion 5-fluorouracil for colorectal cancer: a retrospective efficacy and safety comparison. Clin Colorectal Cancer. 2005 Jul;5(2):89-100. doi: 10.3816/ccc.2005.n.020. PMID 16098249
- [Result] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Result] Taylor FG, Quirke P, Heald RJ, Moran B, Blomqvist L, Swift I, Sebag-Montefiore DJ, Tekkis P, Brown G; MERCURY study group. Preoperative high-resolution magnetic resonance imaging can identify good prognosis stage I, II, and III rectal cancer best managed by surgery alone: a prospective, multicenter, European study. Ann Surg. 2011 Apr;253(4):711-9. doi: 10.1097/SLA.0b013e31820b8d52. PMID 21475011
- [Result] Tiv M, Puyraveau M, Mineur L, Calais G, Maingon P, Bardet E, Mercier M, Bosset JF. Long-term quality of life in patients with rectal cancer treated with preoperative (chemo)-radiotherapy within a randomized trial. Cancer Radiother. 2010 Oct;14(6-7):530-4. doi: 10.1016/j.canrad.2010.06.017. Epub 2010 Aug 24. PMID 20797891
- [Derived] Araujo RO, Vieira FM, Victorino AP, Torres C, Martins I, Guaraldi S, Valadao M, Linhares E, Ferreira CG, Thuler LC. Quality of life in a randomized trial comparing two neoadjuvant regimens for locally advanced rectal cancer-INCAGI004. Support Care Cancer. 2022 Aug;30(8):6557-6572. doi: 10.1007/s00520-022-07059-6. Epub 2022 Apr 29. PMID 35486228